CLINICAL TRIAL: NCT04229940
Title: Randomised Controlled Trial of Peritoneal Bridging Versus no Defect Closure in Laparoscopic Ventral Hernia Repair
Brief Title: Peritoneal in Laparoscopic Ventral Hernia Repair 2
Acronym: BriClo2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Örebro County (Other)
Responsible Party: Principal Investigator, Gabriel Sandblom, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BriClo2
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Hernia, Ventral; Seroma as Procedural Complication
Keywords: Laparoscopy,; Hernia repair
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Intervention Model Description: Double-blind randomized controlled trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient undergoing surgery and the physician performing the follow-up are masked to the allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peritoneal bridging (Experimental): The peritoneum is dissected beginning 2-3 cm from the edge of the defect. The sac is dissected all the way to the opposite edge of the defect. The peritoneal flap is pulled to the opposite side and fixated with Optifix
  Interventions: Procedure: Peritoneal bridging
- No bridging (Active Comparator): The hernia defect is left without closure prior to application of the mesh.
  Interventions: Procedure: No peritoneal bridging

INTERVENTIONS:
Procedure: Peritoneal bridging — The defect is covered by peritoneal bridging
  Arms: Peritoneal bridging
Procedure: No peritoneal bridging — The defect is left without bridging
  Arms: No bridging

SUMMARY:
Laparoscopic ventral hernia repair (VHR) is usually performed by reducing the contents in the hernia sac from the abdominal cavity and then covering the defect from the inside with a mesh, i.e. Intraperitoneal Onlay Mesh (IPOM). This means that the hernia sac is left in situ anterior to the mesh. This may, however, predispose for the development of fluid in the hernia sac, i.e. seroma. The risk of seroma development may be reduced if a the defect is closed before the mesh is applied. Closing the defect may, however, cause tension and pain from the abdominal wall. Instead of closing the defect, the part of the peritoneum constituting the hernia sac may be used for closing the defect. In this case, the peritoneum is dissected from the edges of the hernia sac and then used as a flap that is fixated to the edges of the hernia sac on the opposite side. In a previous study (BriClo), we compared defect closure as control group with peritoneal bridging. That study showed an increased risk for postoperative pain if the defect was closed.

In order to evaluate whether peritoneal bridging reduces the seroma development following ventral hernia repair, we are undertaking a double-blind randomized controlled trial comparing no closure of the defect with peritoneal bridging. The goal is to randomize 100 patients undergoing laparoscopic ventral hernia repair.

Clinical follow-up is performed three months, six months and one year after surgery. At all occasions, the patient is requested to fill in the Ventral Hernia Pain Questionnaire (VHPQ) and an investigation is done in order to assess the presence of seromas, recurrences or other local complications. Duration until return to work is registered. One year after surgery, computer tomography is performed in order to quantify the volume of seromas.

DETAILED DESCRIPTION:
Background Laparoscopic ventral hernia repair (VHR) has become a well-established technique during the last decade. The repair is usually performed by reducing the contents in the hernia sac from the abdominal cavity and then covering the defect from the inside with a mesh, i.e. Intraperitoneal Onlay Mesh (IPOM). This means that the hernia sac is left in situ anterior to the mesh. This may, however, predispose for the development of fluid in the hernia sac, i.e. seroma. Even if the mesh prevents the intestines from protruding into the hernia sac, the patient may still be troubled by discomfort from the seroma that develops in the cavity of the previous hernia sac.

The risk of seroma development may be reduced if a the defect is closed before the mesh is applied (IPOM-Plus). Closing the defect may, however, cause tension and pain from the abdominal wall. Instead of closing the defect, the part of the peritoneum constituting the hernia sac may be used for closing the defect. In this case, the peritoneum is dissected from the edges of the hernia sac and then used as a flap that is fixated to the edges of the hernia sac on the opposite side. This reduces the size of the pseudosac and the peritoneal surface, which prevents transudation to the pseudosac.

In a previous study, we have compared closure of the hernia defect with peritoneal bridging. We found that closure of the defect increased the postoperative pain. In order to assess whether the potential benefit from preitoneal bridging in terms of reduced risk for seromas is present if the defect is not closed, we are undertaking a randomised controlled trial comparing bridging with IPOM without defect closure.

In order to evaluate whether peritoneal bridging reduces the seroma development following ventral hernia repair, we are undertaking a randomized controlled trial. Our goal is to include 50 patients in the study.

Method After obtaining written and oral consent from the patient, the randomisation is performed through a sealed envelope system. The patient is blinded to the allocation. Prior to the procedure, the patient is also requested to fill in the Ventral Hernia Pain Questionnaire (VHPQ).

The procedure is started according to the usual routines. Adhesions covering the defect are dissected to visualize the defect. If the patients is randomized to defect closure, it is sutured with continuous PDS 2-0. In case the patient is allocated to peritoneal bridging, the peritoneum is dissected beginning 2-3 cm from the edge of the defect. The sac is dissected all the way to the opposite edge of the defect. The peritoneal flap is pulled to the opposite side and fixated with Optifix. If the patient is randomized to surgery without bridging, the defect is left without closure.

The mesh is attached in the same, irrespective of randomization. Optifix with double-crown technique is used in both groups. Operation time and intraoperative complications are registered when the procedure is completed. From the day of the procedure until two days postoperatively, pain from the area of surgery is registered daily on a VAS-scale. Time to return to normal daily activities is registered.

The patient is invited to clinical follow-up three months, six months and one year after surgery. At all occasions the patient is requested to fill in VHPQ. One year after surgery, a computer tomography while straining to detect protrusion of the abdominal contents in the defect. Any protrusion seen at the computer tomography is graded according to a previously validated classification. The presence of seromas detected at the computer tomography is described according to Morales-Conde, The computer tomography images are assessed by two radiologists in order to reach consensus. The presence of seroma anterior to the defect is evaluated in terms of size (maximal diameter), localization, shape (round, oval, triangular), mean density (Hounsfield unit, HU) and the volume through three-dimensional reconstructions.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for laparoscopic ventral hernia repair
* Defect size 3-10 cm
* BMI <40

Exclusion Criteria:

* Defect size >10 cm
* Ventral hernias with other localization than the midline
* Emergency surgery and incarcerated hernias
* Preoperative anticipation of extensive adhesions
* Pregnancy or intended pregnancy
* Serious comorbidity (ASA score >3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Seroma volume | One year
  Volume of postoperative seroma measured with ultrasound

SECONDARY OUTCOMES:
Postoperative complications | 30 days
  Complications related to the procedure
Postoperative pain | One year
  Pain assessed with the Ventral Hernia Pain Questionnaire for rating abdominal wall pain. Range 0-7 from no pain to most intensive pain. No subscales or added scores.
Operative time | 3 hours
  Time required to complete the procedure
Hernia recurrence | One year
  Recurrence of the hernia detected clinically or with computer tomography

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Karloskoga Hospital, Karlskoga, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ali F, Sandblom G, Forgo B, Wallin G. Peritoneal Bridging Versus Nonclosure in Laparoscopic Ventral Hernia Repair: A Randomized Controlled Trial. Ann Surg Open. 2023 Feb 2;4(1):e257. doi: 10.1097/AS9.0000000000000257. eCollection 2023 Mar. PMID 37600866